CLINICAL TRIAL: NCT06829459
Title: A Randomized, Controlled, Open-label Phase III Clinical Study to Evaluate the Efficacy and Safety of Glumetinib Combined With Osimertinib Mesylate Versus Platinum-based Doublet Chemotherapy in Non-Small Cell Lung Cancer Patients With MET Amplification and/or Overexpression After Resistance to EGFR-TKIs
Brief Title: A Study to Evaluate the Efficacy and Safety of Glumetinib Combined With Osimertinib Mesylate Versus Platinum-based Doublet Chemotherapy in Non-Small Cell Lung Cancer Patients After Resistance to EGFR-TKIs
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYH2065-002
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — glumetinib; osimertinib; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: Patients those who are eligible for enrollment after screening examinations will be randomized to the investigational group or the control group in a 1:1 ratio by the central randomization system (IWRS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glumetinib combined with osimertinib mesylate (Experimental): Patients will be administered glumetinib 300 mg/dose once daily and osimertinib mesylate 80 mg/dose once daily under fasting conditions in each 21-day treatment cycle. The treatment will continue until IRC-confirmed PD, death, intolerable toxicity, or withdrawal at the patient's discretion (whichever occurs first).
  Interventions: Drug: Glumetinib; Drug: Osimertinib mesylate
- Pemetrexed combined with cisplatin/carboplatin (Active Comparator): Patients will be administered pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2 or carboplatin AUC=5 via intravenous infusion on the first day of each 3-week cycle, for a total of 4 cycles. Patients who have not experienced disease progression (PD) after completing the combination therapy will continue to receive maintenance treatment with pemetrexed following the same regimen until IRC-confirmed PD, death, intolerable toxicity, or withdrawal at the patient's discretion (whichever occurs first). Patients with IRC-confirmed PD may conditionally cross over to receive glumetinib combined with osimertinib at the discretion of the investigator and based on the patient's willingness. The end time of treatment will be determined based on the investigator's assessment of the patient's benefit from participating in the study.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin or carboplatin

INTERVENTIONS:
Drug: Glumetinib — Patients will be administered glumetinib 300 mg/dose once daily once daily under fasting conditions in each 21-day treatment cycle.
  Arms: Glumetinib combined with osimertinib mesylate
Drug: Osimertinib mesylate — Patients will be administered osimertinib mesylate 80 mg/dose once daily under fasting conditions in each 21-day treatment cycle.
  Arms: Glumetinib combined with osimertinib mesylate
Drug: Pemetrexed — Patients will be administered pemetrexed 500 mg/m^2 via intravenous infusion on the first day of each 3-week cycle.
  Arms: Pemetrexed combined with cisplatin/carboplatin
Drug: Cisplatin or carboplatin — Patients will be administered cisplatin 75 mg/m^2 or carboplatin AUC=5 via intravenous infusion on the first day of each 3-week cycle
  Arms: Pemetrexed combined with cisplatin/carboplatin

SUMMARY:
The is a randomized, controlled, open-label Phase III clinical study to evaluate the efficacy and safety of glumetinib combined with osimertinib mesylate versus platinum-based doublet chemotherapy in non-small cell lung cancer( NSCLC) patients with MET amplification and/or overexpression after resistance to EGFR-TKIs..

Approximately 350 NSCLC patients with MET amplification and/or overexpression after previous treatment with EGFR-TKIs are planned to be enrolled. After patients sign the informed consent form (ICF), those who are eligible for enrollment after screening examinations will be randomized to the investigational group or the control group in a 1:1 ratio by the central randomization system (IWRS).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who are able to understand and voluntarily sign the written ICF; 2. Male or female patients aged ≥ 18 years (inclusive); 3. Patients with histologically or cytologically confirmed NSCLC, which is unresectable locally advanced or metastatic (Stage ⅢB, ⅢC, or Ⅳ) NSCLC according to the 8th edition of the TNM Staging System by the International Association for the Study of Lung Cancer (IASLC). Note: If the pathological type is mixed, it should be classified by primary cell type. However, if there are small cell components or neuroendocrine carcinoma components, enrollment will be not allowed; 4. Patients with EGFR-sensitive mutations confirmed by tumor histology or cytology or hematology before the first-line treatment with EGFR-TKIs; 5. Patients who have experienced documented imaging PD after treatment with first-, second- or third-generation EGFR-TKIs (gefitinib, erlotinib, icotinib, afatinib, dacomitinib, osimertinib, etc.); patients who have received prior adjuvant EGFR-TKI treatment after radical surgery may be enrolled if they have had PD within 6 months after the last dose of EGFR-TKIs.

  6. Patients with PD following EGFR-TKI treatment who meet any of the following requirements: a. EGFR T790M negative with MET amplification and/or overexpression after PD following treatment with first- or second-generation EGFR-TKIs; b. MET amplification or overexpression after PD following treatment with third-generation EGFR inhibitors; MET amplification or overexpression in tumor tissue samples as confirmed by the sponsor-designated central laboratory (meeting one of the following conditions):
  1. IHC: 3 +, ≥ 90%
  2. FISH: GCN ≥ 5 or MET/CEP7 ratio ≥ 2 7. Patients who have at least one measurable lesion meeting the RECIST v1.1 criteria. Lesions that have previously undergone local treatments such as radiotherapy can be considered as target lesions upon confirmed progression. Brain metastases will not be considered as target lesions.

     Exclusion Criteria:
* 1. Patients with prior treatment with targeted MET drugs; 2. Patients with T790M-positive mutation after PD following treatment with first- or second-generation EGFR-TKIs; 3. Patients who are positive for other driver genes, such as ALK/ROS1 positive after PD following EGFR-TKI treatment; 4. Patients with prior systemic anti-tumor therapy (including chemotherapy and immunotherapy) for advanced NSCLC other than EGFR-TKIs;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2028-02-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
PFS as assessed by IRC | Up to approximately 24 months after the first patient is enrolled
  Progression-Free-Survival (PFS ) as assessed by IRC

SECONDARY OUTCOMES:
ORR as assessed by IRC | Up to approximately 24 months after the first patient is enrolled
  Objective response rate (ORR) as assessed by IRC
DCRas assessed by IRC | Up to approximately 24 months after the first patient is enrolled
  Disease control rate (DCR) as assessed by IRC
DOR as assessed by IRC | Up to approximately 24 months after the first patient is enrolled
  Duration of response (DOR) as assessed by IRC
OS | Up to approximately 24 months after the first patient is enrolled
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China